CLINICAL TRIAL: NCT03236038
Title: Prevalence of Exocrine Pancreatic Insufficiency in Patients With Decompensated Cirrhosis
Acronym: (EPIIHC)
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Jordi Sanchez-Delgado, M.D; PhD, Corporacion Parc Tauli
Other Study IDs: 2017536
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Exocrine Pancreatic Insufficiency
Keywords: exocrine pancreatic insufficiency; liver cirrhosis; decompensated cirrhosis; malnutrition; prevalence
MeSH Terms: conditions — Exocrine Pancreatic Insufficiency; Liver Cirrhosis; Malnutrition

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Labeled triolein urea breath test — The diagnosis of EPI will be made through the combination of two diagnostic tests.
  The labeled triolein breath test will use criteria established by the manufacturer of the product (Pancreo-Kit®) Isomed pharma.
  The fecal elastase test will be performed at our own center (Bioserv Diagnostics (BS-86-01 Elastase Pancreatic ELISA) distributed by Palex Medical.) In those cases where both results are negative, it will be considered that there is no EPI. In cases where both results are positive, the diagnosis of EPI will be performed. If the results are discordant, a Sobel test or feces quantification test will be performed.
  Other Names: fecal elastase

SUMMARY:
Exocrine pancreatic insufficiency (EPI) is the inability of the pancreas to perform a normal digestive function. The prevalence of IPE in patients with decompensated hepatic cirrhosis (HC) is unknown and most published series are short, old and use a single diagnostic technique with potential risk of false positives and negatives. Demonstrating IPE in a patient with HC can change their vital prognosis with the indication of pancreatic enzymes that can improve their nutritional status and help control their decompensations.

Objectives: To assess the prevalence of IPE in patients with decompensated CH. To establish correlation between fecal elastase and 13C triolein breath test.

Methodology: Unicentric, transversal study that will be carried out during hospitalization. Patients with HC who enter for decompensation and requiere hospitalization will be included consecutively. Exclusion criteria will include prior diagnosis of IPE, suspicion of biliary obstruction, more than 5 dep / d induced by laxatives or liquid stools.

The diagnosis of IPE will be made with the combination of two techniques (13C triolein breath test and fecal elastase).

Demographic, epidemiological data, clinical data as well as anthropometric parameters will be collected. A blood test will also be done to assess nutritional status and associated deficits. A multivariate analysis will be performed to assess the predictive factors of IPE

DETAILED DESCRIPTION:
Exocrine pancreatic insufficiency (EPI) is defined as the inability of the pancreas to perform a normal digestive function. Habitually, it occurs as a result of a severe reduction in the secretion of pancreatic enzymes, although - less frequently - it may be due to the inability of these enzymes to perform their function. Clinically, it has a very broad spectrum of presentation with abdominal discomforts, malnutrition, chronic diarrhea and, in severe cases, steatorrhea. It must be said, however, that it is not until the disease is very evolved with a pancreatic function very deteriorated (more than 90%) that steatorrhea becomes clinically evident. In addition, the onset of symptoms triggered by the intake of fats makes these patients adapt their diet, often unconsciously, so it is not uncommon to find patients with EPI and constipation.

To establish the diagnosis of IPE, different clinical tests are used. There are direct methods or invasive (secretin stimulation test, secretin-cerulein Lundh test) and noninvasive or indirect methods (coefficient of fat absorption, fecal elastase, fecal chymotrypsin activity, the pancreoleuril test, test with paraaminobenzoic acid and marked triolein test) are, in general, more accessible to the usual clinical practice.

Regarding etiology, the most frequent cause of EPI is chronic pancreatitis, an entity that is closely linked to chronic alcohol consumption. On the one hand, it should be noted that alcohol is a common etiologic factor to both pathogenesis of pancreatic and liver affections. On the other hand, it is well known that the liver and pancreas have a close relationship with regard to their anatomy and physiology. The pancreatic duct and the coledocus bind to the level of the Vater papilla, so that their contents are mixed.

Patients with EPI have severe malnutrition, a factor which increases the morbidity and mortality. Therefore, adequately replacing nutritional deficits by enzyme replacement therapy contributes significantly to decrease the complications, the hospital stays and the mortality. It could increase the quality of life of the patients. In addition, patients suffering from liver cirrhosis have other complications arising from malnutrition, as ascites that could be benefited from the improvement of the nutritional profile by enzyme replacement therapy detected in case of EPI. That is why we believe that our study could contribute to improving patient management with decompensated liver cirrhosis.

The objective of the study is to assess the prevalence of exocrine pancreatic insufficiency EPI in patients with decompensated alcoholic liver cirrhosis.

This is an epidemiological, unicentral, cross-sectional study that will be carried out within the hospital setting from October '17 to October'19.

Patients diagnosed with liver cirrrhosis and enter the hepatology unit for clinical decompensation (sd hepatorenal, ascitic decompensation, hepatic encephalopathy, gastrointestinal bleeding stable) will be included .

The investigators will collect demographic, epidemiology, analytic and clinical data. Anthropometric parameters such as tricipital fold, weight and size, will also be measured, which will allow the calculation of body mass index (BMI).

In order to diagnose the presence of IPE, the breath test with triolein marked with 13C (Pancreo-Kit®) will be performed. The study consists of a delay of 8 hours (overnight) and later obtaining a basal sample through exhalation of air in a tube. Subsequently, a substrate (foods with marked triolein) will be administered to the patient and after 30 minutes, it will have to exhale air in a tube every 30 minutes for a total of 6 hours, thus obtaining a total of 13 samples.

Blood tests will also be performed on all patients to assess their nutritional status (Hg, albumin, prealbumin, total proteins, cholesterol (HDL / LDL), bilirubin, prothrombin time, triglycerides, liposoluble Vitamins A, D, E and K; Vitamins B1, B12; calcium, phosphorus and magnesium), Hb glucose and collect a sample of solid stool isolated for the determination of the fecal elastase.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histological diagnosis of CH or by clinical, analytical, ecographic or fibroscan criteria.
2. Patients with decompensated HC (ascites, hepatic hydrothorax, hepatorenal syndrome, digestive bleeding due to portal hypertension or hepatic encephalopathy.
3. Signature of informed consent
4. Prevision of hospital admission for a minimum of 48 hours (for the correct completion of the marked triolein test and the collection of samples for fecal elastase)
5. Age between 18 and 85 years.

Exclusion Criteria:

1. Previous diagnosis of EPI
2. Suspected biliary tract obstruction
3. Need for high doses of laxative which makes it impossible to collect faecal samples correctly (> 5 dep / d secondary to laxatives)
4. Patients who, due to their clinical situation, are unable to collaborate in the labeled triolein breath test
5. Patients with inability to use the oral route.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with decompensated liver cirrhosis and who are admitted to hospital for this reason. Patients will be included prospectively and consecutively.
Sampling Method: Non-Probability Sample
Enrollment: 125 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-01 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of exocrine pancreatic insufficiency in decompensated alcoholic cirrhosis | This is a prevalence study. Outcome measure will be assessed during patient admision in the hospital. Data will be reported once the inclusion has been completed (2 years).
  The diagnosis of EPI will be made through the combination of two diagnostic tests.
  The labeled triolein breath test will use criteria established by the manufacturer of the product (Pancreo-Kit®) Isomed pharma.
  Reference value: Normal: > 29%; Pathological: < 29% of the fat administered
  The fecal elastase test (Bioserv Diagnostics (BS-86-01 Elastase Pancreatic ELISA) distributed by Palex Medical.)
  * A normal result will be considered: 200 to > 500 μg / g
  * Slight exocrine pancreatic insufficiency- Moderate: 100 - 200 μg / g
  * Severe exocrine pancreatic insufficiency: <100 μg / g
  In those cases where both results are negative, it will be considered that there is no EPI. In cases where both results are positive, the diagnosis of EPI will be performed. If the results are discordant, a Sobel test or feces quantification test will be performed.
  Coefficient of fat absorption; Pathological if elimination > 7g of fat / day with a diet of 100g fat / day.

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Sánchez-Delgado, M.D; PhD, Principal Investigator — Corporació Sanitària Parc Tauli
Locations (1):
- Parc Tauli Hospital, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Aoufi Rabih S, Garcia Agudo R, Legaz Huidobro ML, Ynfante Ferrus M, Gonzalez Carro P, Perez Roldan F, Ruiz Carrillo F, Tenias Burillo JM. Exocrine pancreatic insufficiency and chronic pancreatitis in chronic alcoholic liver disease: coincidence or shared toxicity? Pancreas. 2014 Jul;43(5):730-4. doi: 10.1097/MPA.0000000000000085. PMID 24713840